CLINICAL TRIAL: NCT00005152
Title: Nurses' Health Study (Cardiovascular Component)
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, JoAnn E. Manson, MD, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2008P000327; R01HL034594-28 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Coronary Disease; Heart Diseases; Cerebrovascular Accident; Pulmonary Embolism; Angina Pectoris; Myocardial Infarction; Menopause; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Coronary Disease; Heart Diseases; Stroke; Pulmonary Embolism; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the relationships of hormonal, reproductive, dietary, and lifestyle factors, as well as biochemical and genetic factors, with the subsequent risk of coronary heart disease and other cardiovascular events in a cohort of female registered nurses. The current funding cycle involves comprehensive metabolomic profiling of coronary heart disease cases and controls and development of metabolomic risk scores for coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The Nurses' Health Study began in 1976, when 121,700 female registered nurses living in eleven states completed a mailed questionnaire that included items about their medical history, diet, and other risk factors for cancer. The National Cancer Institute funded the first three years of the study and subsequent years on data pertaining to cancer. In 1980 the National Heart, Lung, and Blood Institute began funding the cardiovascular portion of the study. Follow-up questionnaires have been administered every two years subsequently. Blood samples were collected on a subsample of the women between 1989-1990 and stored for analysis of germline DNA and circulating biomarkers.

The cardiovascular component is funded through May 2029.

DESIGN NARRATIVE:

In 1976, 121,700 nurses ages 30-55 completed and returned the initial Nurses' Health Study questionnaire and comprise the Nurses' Health Study cohort. The cohort has been followed by means of biennial mailed questionnaires. A total of 109,413 participants responded to the 1978 questionnaire. In addition, 400 women who replied in 1976 stated that they did not wish to continue in the study and 390 women died. In 1980, the first major dietary assessment was added to the questionnaire. In the 1978-1980 interval, there were 624 deaths, 300 women declined further participation, approximately 99,000 completed the full questionnaire including the dietary questionnaire, and another 4,000 completed an abbreviated questionnaire, for a total of about 103,000 responses. In 1982, the overall response was 101,174. The approximately 19,000 living non-respondents were followed by telephone, yielding 71 percent of the non-respondents. Thus, at the end of 1982, current information was available on 116,150 or 95.4 percent of the original cohort. A subset of 32,826 women provided blood samples between 1989 and 1990. Genotyping on 1,186 women (382 with coronary heart disease and 804 matched controls) was performed using Affymetrix 6.0 platform.

Deaths in the cohort were usually reported by next-of-kin or postal authorities. At the completion of each mailing cycle, the National Death Index was searched for names of non-respondents who might have died. By comparing deaths ascertained from independent sources, the study ascertained an estimated 98 percent of deaths. Death certificates were obtained from state vital statistics departments to confirm all reported deaths. For all death certificates indicating possible cardiovascular disease, permission to obtain further information was requested from family members. Confirmed coronary heart disease death required additional information beyond the death certificate such as autopsy reports, ECG and enzyme changes of myocardial infarction prior to death, classical chest pain immediately prior to death, prior documented myocardial infarction or angina, or prior cardiac catheterization showing severe coronary disease.

Data were collected on date of birth, weight, cigarette smoking, menopausal status and current interim use of menopausal hormone therapy. Data were also collected on incident cases of nonfatal myocardial infarction, stroke, pulmonary embolism, and angina pectoris. These items appeared on each questionnaire. In addition, nutritional parameters were assessed by a self-administered semi-quantitative food frequency questionnaire in 1986 and again in 1990.

The study was renewed in 1993 with particular attention given to dietary antioxidants, other nutritional factors, physical activity, regional fat distribution, menopausal estrogen and progestin therapy, and biochemical markers including plasma lipids and apoproteins. Follow-up for nonfatal cardiovascular disease events is over 92 percent for the original 121,700 participants. Fatal cardiovascular events are documented by death certificates and confirmed and classified by review of hospital records, autopsy reports, and interviews with next of kin. Searches of the National Death Index for all nonrespondents ensure the identification of remaining deaths, resulting in mortality follow-up that is more than 98 percent complete.

The study was renewed in FY 2002 to continue follow-up through March 2007. A major aim of that renewal was to compare the predictive capability of several biochemical and genetic markers of inflammation and endothelial activation for coronary heart disease versus stroke in women: C-reactive protein (CRP), E-selectin, intercellular adhesion molecule-1, endothelin-1, and polymorphisms of the CRP and E-selectin genes. The study also continues the investigation of lifestyle determinants of cardiovascular disease, including menopausal hormone therapy (dose, formulation, and duration of use) and alcohol consumption (dose and beverage type), in the full cohort, and interactions of these exposures with the above biomarkers and with novel genetic markers (prothrombin and alcohol dehydrogenase-3 gene polymorphisms). Genotypes from 1,186 women typed as part of a genome-wide association study of coronary heart disease were used to study genetic factors associated with cardiovascular disease and the interplay of genes and diet on cardiovascular risk. Subsequent renewal cycles included study of plasma adipokines and metabolomic predictors, including gut flora metabolites such as trimethylamine N-oxide, choline, and L-carnitine, of coronary heart disease; and comprehensive metabolomic profiling of coronary heart disease cases and controls and development of metabolomic risk scores for coronary heart disease. During the current funding cycle, researchers will conduct comprehensive proteomic profiling of coronary heart disease risk and the relationship to diet and other lifestyle factors.

ELIGIBILITY:
See "Detailed Description"

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: See "Detailed Description"
Sampling Method: Probability Sample
Enrollment: 121700 (Actual)
Dates: Start 1980-08; Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Coronary heart disease (CHD) | The primary outcome measure time frame is first CHD event during person-time of follow-up for each participant from study enrollment through March 2022.
  CHD is defined as nonfatal myocardial infarction and death from coronary heart disease. Information on the outcome is assessed by medical record review of events reported on biennial questionnaires or by searches of the National Death Index, and the date of the CHD event or CHD death is ascertained from these sources.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn E Manson, MD, DrPH, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Background] Willett WC, Hennekens CH, Bain C, Rosner B, Speizer FE. Cigarette smoking and non-fatal myocardial infarction in women. Am J Epidemiol. 1981 May;113(5):575-82. doi: 10.1093/oxfordjournals.aje.a113134. PMID 7223737
- [Background] Bain C, Willett W, Hennekens CH, Rosner B, Belanger C, Speizer FE. Use of postmenopausal hormones and risk of myocardial infarction. Circulation. 1981 Jul;64(1):42-6. doi: 10.1161/01.cir.64.1.42. PMID 7237723
- [Background] Rosenberg L, Hennekens CH, Rosner B, Belanger C, Rothman KJ, Speizer FE. Early menopause and the risk of myocardial infarction. Am J Obstet Gynecol. 1981 Jan;139(1):47-51. doi: 10.1016/0002-9378(81)90410-5. PMID 7457520
- [Background] Willett W, Stampfer MJ, Bain C, Lipnick R, Speizer FE, Rosner B, Cramer D, Hennekens CH. Cigarette smoking, relative weight, and menopause. Am J Epidemiol. 1983 Jun;117(6):651-8. doi: 10.1093/oxfordjournals.aje.a113598. PMID 6859020
- [Background] Stampfer MJ, Willett WC, Speizer FE, Dysert DC, Lipnick R, Rosner B, Hennekens CH. Test of the National Death Index. Am J Epidemiol. 1984 May;119(5):837-9. doi: 10.1093/oxfordjournals.aje.a113804. No abstract available. PMID 6720679
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201
- [Background] Stampfer MJ, Willett WC, Colditz GA, Rosner B, Speizer FE, Hennekens CH. A prospective study of postmenopausal estrogen therapy and coronary heart disease. N Engl J Med. 1985 Oct 24;313(17):1044-9. doi: 10.1056/NEJM198510243131703. PMID 4047106
- [Background] Colditz GA, Stampfer MJ, Willett WC, Rosner B, Speizer FE, Hennekens CH. A prospective study of parental history of myocardial infarction and coronary heart disease in women. Am J Epidemiol. 1986 Jan;123(1):48-58. doi: 10.1093/oxfordjournals.aje.a114223. PMID 3940442
- [Background] Colditz GA, Martin P, Stampfer MJ, Willett WC, Sampson L, Rosner B, Hennekens CH, Speizer FE. Validation of questionnaire information on risk factors and disease outcomes in a prospective cohort study of women. Am J Epidemiol. 1986 May;123(5):894-900. doi: 10.1093/oxfordjournals.aje.a114319. PMID 3962971
- [Background] Colditz GA, Willett WC, Stampfer MJ, Rosner B, Speizer FE, Hennekens CH. Menopause and the risk of coronary heart disease in women. N Engl J Med. 1987 Apr 30;316(18):1105-10. doi: 10.1056/NEJM198704303161801. PMID 3574358
- [Background] Colditz GA, Willett WC, Stampfer MJ, Rosner B, Speizer FE, Hennekens CH. A prospective study of age at menarche, parity, age at first birth, and coronary heart disease in women. Am J Epidemiol. 1987 Nov;126(5):861-70. doi: 10.1093/oxfordjournals.aje.a114723. PMID 3661534
- [Background] Willett WC, Green A, Stampfer MJ, Speizer FE, Colditz GA, Rosner B, Monson RR, Stason W, Hennekens CH. Relative and absolute excess risks of coronary heart disease among women who smoke cigarettes. N Engl J Med. 1987 Nov 19;317(21):1303-9. doi: 10.1056/NEJM198711193172102. PMID 3683458
- [Background] Colditz GA, Willett WC, Stampfer MJ, Sampson L, Rosner B, Hennekens CH, Speizer FE. The influence of age, relative weight, smoking, and alcohol intake on the reproducibility of a dietary questionnaire. Int J Epidemiol. 1987 Sep;16(3):392-8. doi: 10.1093/ije/16.3.392. PMID 3667037
- [Background] Stampfer MJ, Colditz GA, Willett WC, Rosner B, Speizer FE, Hennekens CH: Coronary Risk Factors in Women - the Nurses' Health Study Experience. In: Proceedings of an NIH Workshop on Coronary Heart Disease in Women, Eaker ED, Packard B, Wenger NK et al (Eds). Haymarket Doyma, Inc. New York, 1987
- [Background] Willett WC, Sampson L, Browne ML, Stampfer MJ, Rosner B, Hennekens CH, Speizer FE. The use of a self-administered questionnaire to assess diet four years in the past. Am J Epidemiol. 1988 Jan;127(1):188-99. doi: 10.1093/oxfordjournals.aje.a114780. PMID 3337073
- [Background] Romieu I, Willett WC, Stampfer MJ, Colditz GA, Sampson L, Rosner B, Hennekens CH, Speizer FE. Energy intake and other determinants of relative weight. Am J Clin Nutr. 1988 Mar;47(3):406-12. doi: 10.1093/ajcn/47.3.406. PMID 3348153
- [Background] Colditz GA, Bonita R, Stampfer MJ, Willett WC, Rosner B, Speizer FE, Hennekens CH. Cigarette smoking and risk of stroke in middle-aged women. N Engl J Med. 1988 Apr 14;318(15):937-41. doi: 10.1056/NEJM198804143181501. PMID 3352685
- [Background] Stampfer MJ, Colditz GA, Willett WC, Speizer FE, Hennekens CH. A prospective study of moderate alcohol consumption and the risk of coronary disease and stroke in women. N Engl J Med. 1988 Aug 4;319(5):267-73. doi: 10.1056/NEJM198808043190503. PMID 3393181
- [Background] Stampfer MJ, Colditz GA, Willett WC, Manson JE, Arky RA, Hennekens CH, Speizer FE. A prospective study of moderate alcohol drinking and risk of diabetes in women. Am J Epidemiol. 1988 Sep;128(3):549-58. doi: 10.1093/oxfordjournals.aje.a115002. PMID 3414660
- [Background] Stampfer MJ, Willett WC, Colditz GA, Speizer FE, Hennekens CH. A prospective study of past use of oral contraceptive agents and risk of cardiovascular diseases. N Engl J Med. 1988 Nov 17;319(20):1313-7. doi: 10.1056/NEJM198811173192004. PMID 3185634
- [Background] Fiebach NH, Hebert PR, Stampfer MJ, Colditz GA, Willett WC, Rosner B, Speizer FE, Hennekens CH. A prospective study of high blood pressure and cardiovascular disease in women. Am J Epidemiol. 1989 Oct;130(4):646-54. doi: 10.1093/oxfordjournals.aje.a115386. PMID 2773913
- [Background] Witteman JC, Willett WC, Stampfer MJ, Colditz GA, Sacks FM, Speizer FE, Rosner B, Hennekens CH. A prospective study of nutritional factors and hypertension among US women. Circulation. 1989 Nov;80(5):1320-7. doi: 10.1161/01.cir.80.5.1320. PMID 2805268
- [Background] Witteman JC, Willett WC, Stampfer MJ, Colditz GA, Kok FJ, Sacks FM, Speizer FE, Rosner B, Hennekens CH. Relation of moderate alcohol consumption and risk of systemic hypertension in women. Am J Cardiol. 1990 Mar 1;65(9):633-7. doi: 10.1016/0002-9149(90)91043-6. PMID 2309634
- [Background] Manson JE, Colditz GA, Stampfer MJ, Willett WC, Rosner B, Monson RR, Speizer FE, Hennekens CH. A prospective study of obesity and risk of coronary heart disease in women. N Engl J Med. 1990 Mar 29;322(13):882-9. doi: 10.1056/NEJM199003293221303. PMID 2314422
- [Background] Stampfer MJ, Willett WC, Colditz GA, Speizer FE, Hennekens CH. Past use of oral contraceptives and cardiovascular disease: a meta-analysis in the context of the Nurses' Health Study. Am J Obstet Gynecol. 1990 Jul;163(1 Pt 2):285-91. doi: 10.1016/0002-9378(90)90569-s. PMID 2142573
- [Background] Manson JE, Rimm EB, Colditz GA, Willett WC, Nathan DM, Arky RA, Rosner B, Hennekens CH, Speizer FE, Stampfer MJ. A prospective study of postmenopausal estrogen therapy and subsequent incidence of non-insulin-dependent diabetes mellitus. Ann Epidemiol. 1992 Sep;2(5):665-73. doi: 10.1016/1047-2797(92)90011-e. PMID 1342318
- [Background] Manson JE, Rimm EB, Colditz GA, Stampfer MJ, Willett WC, Arky RA, Rosner B, Hennekens CH, Speizer FE. Parity and incidence of non-insulin-dependent diabetes mellitus. Am J Med. 1992 Jul;93(1):13-8. doi: 10.1016/0002-9343(92)90674-z. PMID 1626567
- [Background] Colditz GA. A prospective assessment of moderate alcohol intake and major chronic diseases. Ann Epidemiol. 1990 Dec;1(2):167-77. doi: 10.1016/1047-2797(90)90007-f. PMID 1669497
- [Background] Manson JE, Stampfer MJ, Colditz GA, Willett WC, Rosner B, Speizer FE, Hennekens CH. A prospective study of aspirin use and primary prevention of cardiovascular disease in women. JAMA. 1991 Jul 24-31;266(4):521-7. PMID 2061978
- [Background] Manson JE, Colditz GA, Stampfer MJ, Willett WC, Krolewski AS, Rosner B, Arky RA, Speizer FE, Hennekens CH. A prospective study of maturity-onset diabetes mellitus and risk of coronary heart disease and stroke in women. Arch Intern Med. 1991 Jun;151(6):1141-7. PMID 2043016
- [Background] Kawachi I, Colditz GA, Stampfer MJ, Willett WC, Manson JE, Speizer FE, Hennekens CH. Prospective study of shift work and risk of coronary heart disease in women. Circulation. 1995 Dec 1;92(11):3178-82. doi: 10.1161/01.cir.92.11.3178. PMID 7586301
- [Background] Willett WC, Manson JE, Stampfer MJ, Colditz GA, Rosner B, Speizer FE, Hennekens CH. Weight, weight change, and coronary heart disease in women. Risk within the 'normal' weight range. JAMA. 1995 Feb 8;273(6):461-5. doi: 10.1001/jama.1995.03520300035033. PMID 7654270
- [Background] Gliksman MD, Kawachi I, Hunter D, Colditz GA, Manson JE, Stampfer MJ, Speizer FE, Willett WC, Hennekens CH. Childhood socioeconomic status and risk of cardiovascular disease in middle aged US women: a prospective study. J Epidemiol Community Health. 1995 Feb;49(1):10-5. doi: 10.1136/jech.49.1.10. PMID 7706992
- [Background] Manson JE. Postmenopausal hormone therapy and atherosclerotic disease. Am Heart J. 1994 Dec;128(6 Pt 2):1337-43. doi: 10.1016/0002-8703(94)90257-7. PMID 7977016
- [Background] Manson JE, Spelsberg A. Primary prevention of non-insulin-dependent diabetes mellitus. Am J Prev Med. 1994 May-Jun;10(3):172-84. PMID 7917445
- [Background] Kawachi I, Colditz GA, Stampfer MJ, Willett WC, Manson JE, Rosner B, Hunter DJ, Hennekens CH, Speizer FE. Smoking cessation in relation to total mortality rates in women. A prospective cohort study. Ann Intern Med. 1993 Nov 15;119(10):992-1000. doi: 10.7326/0003-4819-119-10-199311150-00005. PMID 8214996
- [Background] Rich-Edwards JW, Manson JE, Stampfer MJ, Colditz GA, Willett WC, Rosner B, Speizer FE, Hennekens CH. Height and the risk of cardiovascular disease in women. Am J Epidemiol. 1995 Nov 1;142(9):909-17. doi: 10.1093/oxfordjournals.aje.a117738. PMID 7572971
- [Background] Rich-Edwards JW, Stampfer MJ, Manson JE, Rosner B, Hankinson SE, Colditz GA, Willett WC, Hennekens CH. Birth weight and risk of cardiovascular disease in a cohort of women followed up since 1976. BMJ. 1997 Aug 16;315(7105):396-400. doi: 10.1136/bmj.315.7105.396. PMID 9277603
- [Background] Kawachi I, Colditz GA, Speizer FE, Manson JE, Stampfer MJ, Willett WC, Hennekens CH. A prospective study of passive smoking and coronary heart disease. Circulation. 1997 May 20;95(10):2374-9. doi: 10.1161/01.cir.95.10.2374. PMID 9170399
- [Background] Goldhaber SZ, Grodstein F, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Willett WC, Hennekens CH. A prospective study of risk factors for pulmonary embolism in women. JAMA. 1997 Feb 26;277(8):642-5. PMID 9039882
- [Background] Grodstein F, Stampfer MJ, Goldhaber SZ, Manson JE, Colditz GA, Speizer FE, Willett WC, Hennekens CH. Prospective study of exogenous hormones and risk of pulmonary embolism in women. Lancet. 1996 Oct 12;348(9033):983-7. doi: 10.1016/S0140-6736(96)07308-4. PMID 8855854
- [Background] Willett WC, Stampfer MJ, Manson JE, Colditz GA, Rosner BA, Speizer FE, Hennekens CH. Coffee consumption and coronary heart disease in women. A ten-year follow-up. JAMA. 1996 Feb 14;275(6):458-62. doi: 10.1001/jama.1996.03530300042038. PMID 8627967
- [Background] Ascherio A, Hennekens C, Willett WC, Sacks F, Rosner B, Manson J, Witteman J, Stampfer MJ. Prospective study of nutritional factors, blood pressure, and hypertension among US women. Hypertension. 1996 May;27(5):1065-72. doi: 10.1161/01.hyp.27.5.1065. PMID 8621198
- [Background] Kawachi I, Willett WC, Colditz GA, Stampfer MJ, Speizer FE. A prospective study of coffee drinking and suicide in women. Arch Intern Med. 1996 Mar 11;156(5):521-5. PMID 8604958
- [Background] Califf RM, Kramer JM. What have we learned from the calcium channel blocker controversy? Circulation. 1998 Apr 28;97(16):1529-31. doi: 10.1161/01.cir.97.16.1529. No abstract available. PMID 9593555
- [Background] Hu FB, Willett WC, Manson JE, Colditz GA, Rimm EB, Speizer FE, Hennekens CH, Stampfer MJ. Snoring and risk of cardiovascular disease in women. J Am Coll Cardiol. 2000 Feb;35(2):308-13. doi: 10.1016/s0735-1097(99)00540-9. PMID 10676674
- [Background] Michels KB, Rosner BA, Manson JE, Stampfer MJ, Walker AM, Willett WC, Hennekens CH. Prospective study of calcium channel blocker use, cardiovascular disease, and total mortality among hypertensive women: the Nurses' Health Study. Circulation. 1998 Apr 28;97(16):1540-8. doi: 10.1161/01.cir.97.16.1540. PMID 9593558
- [Background] Rimm EB, Willett WC, Hu FB, Sampson L, Colditz GA, Manson JE, Hennekens C, Stampfer MJ. Folate and vitamin B6 from diet and supplements in relation to risk of coronary heart disease among women. JAMA. 1998 Feb 4;279(5):359-64. doi: 10.1001/jama.279.5.359. PMID 9459468
- [Background] Rexrode KM, Hennekens CH, Willett WC, Colditz GA, Stampfer MJ, Rich-Edwards JW, Speizer FE, Manson JE. A prospective study of body mass index, weight change, and risk of stroke in women. JAMA. 1997 May 21;277(19):1539-45. doi: 10.1001/jama.1997.03540430051032. PMID 9153368
- [Background] Iso H, Rexrode K, Hennekens CH, Manson JE. Application of computer tomography-oriented criteria for stroke subtype classification in a prospective study. Ann Epidemiol. 2000 Feb;10(2):81-7. doi: 10.1016/s1047-2797(99)00040-x. PMID 10691061
- [Background] Fine JT, Colditz GA, Coakley EH, Moseley G, Manson JE, Willett WC, Kawachi I. A prospective study of weight change and health-related quality of life in women. JAMA. 1999 Dec 8;282(22):2136-42. doi: 10.1001/jama.282.22.2136. PMID 10591335
- [Background] Hu FB, Stampfer MJ, Manson JE, Ascherio A, Colditz GA, Speizer FE, Hennekens CH, Willett WC. Dietary saturated fats and their food sources in relation to the risk of coronary heart disease in women. Am J Clin Nutr. 1999 Dec;70(6):1001-8. doi: 10.1093/ajcn/70.6.1001. PMID 10584044
- [Background] Hu FB, Willett WC, Colditz GA, Ascherio A, Speizer FE, Rosner B, Hennekens CH, Stampfer MJ. Prospective study of snoring and risk of hypertension in women. Am J Epidemiol. 1999 Oct 15;150(8):806-16. doi: 10.1093/oxfordjournals.aje.a010085. PMID 10522651
- [Background] Liu S, Stampfer MJ, Hu FB, Giovannucci E, Rimm E, Manson JE, Hennekens CH, Willett WC. Whole-grain consumption and risk of coronary heart disease: results from the Nurses' Health Study. Am J Clin Nutr. 1999 Sep;70(3):412-9. doi: 10.1093/ajcn/70.3.412. PMID 10479204
- [Background] Iso H, Stampfer MJ, Manson JE, Rexrode K, Hennekens CH, Colditz GA, Speizer FE, Willett WC. Prospective study of calcium, potassium, and magnesium intake and risk of stroke in women. Stroke. 1999 Sep;30(9):1772-9. doi: 10.1161/01.str.30.9.1772. PMID 10471422
- [Background] Iso H, Hennekens CH, Stampfer MJ, Rexrode KM, Colditz GA, Speizer FE, Willett WC, Manson JE. Prospective study of aspirin use and risk of stroke in women. Stroke. 1999 Sep;30(9):1764-71. doi: 10.1161/01.str.30.9.1764. PMID 10471421
- [Background] Manson JE, Hu FB, Rich-Edwards JW, Colditz GA, Stampfer MJ, Willett WC, Speizer FE, Hennekens CH. A prospective study of walking as compared with vigorous exercise in the prevention of coronary heart disease in women. N Engl J Med. 1999 Aug 26;341(9):650-8. doi: 10.1056/NEJM199908263410904. PMID 10460816
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm E, Colditz GA, Speizer FE, Hennekens CH, Willett WC. Dietary protein and risk of ischemic heart disease in women. Am J Clin Nutr. 1999 Aug;70(2):221-7. doi: 10.1093/ajcn.70.2.221. PMID 10426698
- [Background] Hu FB, Grodstein F, Hennekens CH, Colditz GA, Johnson M, Manson JE, Rosner B, Stampfer MJ. Age at natural menopause and risk of cardiovascular disease. Arch Intern Med. 1999 May 24;159(10):1061-6. doi: 10.1001/archinte.159.10.1061. PMID 10335682
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm EB, Wolk A, Colditz GA, Hennekens CH, Willett WC. Dietary intake of alpha-linolenic acid and risk of fatal ischemic heart disease among women. Am J Clin Nutr. 1999 May;69(5):890-7. doi: 10.1093/ajcn/69.5.890. PMID 10232627
- [Background] Cornuz J, Feskanich D, Willett WC, Colditz GA. Smoking, smoking cessation, and risk of hip fracture in women. Am J Med. 1999 Mar;106(3):311-4. doi: 10.1016/s0002-9343(99)00022-4. PMID 10190380
- [Background] Hu FB, Stampfer MJ, Rimm E, Ascherio A, Rosner BA, Spiegelman D, Willett WC. Dietary fat and coronary heart disease: a comparison of approaches for adjusting for total energy intake and modeling repeated dietary measurements. Am J Epidemiol. 1999 Mar 15;149(6):531-40. doi: 10.1093/oxfordjournals.aje.a009849. PMID 10084242
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm EB, Colditz GA, Rosner BA, Speizer FE, Hennekens CH, Willett WC. Frequent nut consumption and risk of coronary heart disease in women: prospective cohort study. BMJ. 1998 Nov 14;317(7169):1341-5. doi: 10.1136/bmj.317.7169.1341. PMID 9812929
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm E, Colditz GA, Rosner BA, Hennekens CH, Willett WC. Dietary fat intake and the risk of coronary heart disease in women. N Engl J Med. 1997 Nov 20;337(21):1491-9. doi: 10.1056/NEJM199711203372102. PMID 9366580
- [Background] Hu FB, Stampfer MJ, Colditz GA, Ascherio A, Rexrode KM, Willett WC, Manson JE. Physical activity and risk of stroke in women. JAMA. 2000 Jun 14;283(22):2961-7. doi: 10.1001/jama.283.22.2961. PMID 10865274
- [Background] Stampfer MJ, Hu FB, Manson JE, Rimm EB, Willett WC. Primary prevention of coronary heart disease in women through diet and lifestyle. N Engl J Med. 2000 Jul 6;343(1):16-22. doi: 10.1056/NEJM200007063430103. PMID 10882764
- [Background] Solomon CG, Hu FB, Stampfer MJ, Colditz GA, Speizer FE, Rimm EB, Willett WC, Manson JE. Moderate alcohol consumption and risk of coronary heart disease among women with type 2 diabetes mellitus. Circulation. 2000 Aug 1;102(5):494-9. doi: 10.1161/01.cir.102.5.494. PMID 10920059
- [Background] Liu S, Manson JE, Stampfer MJ, Rexrode KM, Hu FB, Rimm EB, Willett WC. Whole grain consumption and risk of ischemic stroke in women: A prospective study. JAMA. 2000 Sep 27;284(12):1534-40. doi: 10.1001/jama.284.12.1534. PMID 11000647
- [Background] Hu FB, Stampfer MJ, Manson JE, Grodstein F, Colditz GA, Speizer FE, Willett WC. Trends in the incidence of coronary heart disease and changes in diet and lifestyle in women. N Engl J Med. 2000 Aug 24;343(8):530-7. doi: 10.1056/NEJM200008243430802. PMID 10954760
- [Background] Iso H, Rexrode KM, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Hennekens CH, Willett WC. Intake of fish and omega-3 fatty acids and risk of stroke in women. JAMA. 2001 Jan 17;285(3):304-12. doi: 10.1001/jama.285.3.304. PMID 11176840
- [Background] Hu FB, Hankinson SE, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Hennekens CH, Willett WC. Prospective study of cataract extraction and risk of coronary heart disease in women. Am J Epidemiol. 2001 May 1;153(9):875-81. doi: 10.1093/aje/153.9.875. PMID 11323318
- [Background] Liu S, Manson JE, Stampfer MJ, Holmes MD, Hu FB, Hankinson SE, Willett WC. Dietary glycemic load assessed by food-frequency questionnaire in relation to plasma high-density-lipoprotein cholesterol and fasting plasma triacylglycerols in postmenopausal women. Am J Clin Nutr. 2001 Mar;73(3):560-6. doi: 10.1093/ajcn/73.3.560. PMID 11237932
- [Background] Iso H, Stampfer MJ, Manson JE, Rexrode K, Hu F, Hennekens CH, Colditz GA, Speizer FE, Willett WC. Prospective study of fat and protein intake and risk of intraparenchymal hemorrhage in women. Circulation. 2001 Feb 13;103(6):856-63. doi: 10.1161/01.cir.103.6.856. PMID 11171795
- [Background] Joshipura KJ, Hu FB, Manson JE, Stampfer MJ, Rimm EB, Speizer FE, Colditz G, Ascherio A, Rosner B, Spiegelman D, Willett WC. The effect of fruit and vegetable intake on risk for coronary heart disease. Ann Intern Med. 2001 Jun 19;134(12):1106-14. doi: 10.7326/0003-4819-134-12-200106190-00010. PMID 11412050
- [Background] Al-Delaimy WK, Manson JE, Solomon CG, Kawachi I, Stampfer MJ, Willett WC, Hu FB. Smoking and risk of coronary heart disease among women with type 2 diabetes mellitus. Arch Intern Med. 2002 Feb 11;162(3):273-9. doi: 10.1001/archinte.162.3.273. PMID 11822919
- [Background] Fung TT, Willett WC, Stampfer MJ, Manson JE, Hu FB. Dietary patterns and the risk of coronary heart disease in women. Arch Intern Med. 2001 Aug 13-27;161(15):1857-62. doi: 10.1001/archinte.161.15.1857. PMID 11493127
- [Background] Hu FB, Stampfer MJ, Solomon CG, Liu S, Willett WC, Speizer FE, Nathan DM, Manson JE. The impact of diabetes mellitus on mortality from all causes and coronary heart disease in women: 20 years of follow-up. Arch Intern Med. 2001 Jul 23;161(14):1717-23. doi: 10.1001/archinte.161.14.1717. PMID 11485504
- [Background] Hu FB, Willett WC. Diet and coronary heart disease: findings from the Nurses' Health Study and Health Professionals' Follow-up Study. J Nutr Health Aging. 2001;5(3):132-8. PMID 11458281
- [Background] Grodstein F, Manson JE, Stampfer MJ. Postmenopausal hormone use and secondary prevention of coronary events in the nurses' health study. a prospective, observational study. Ann Intern Med. 2001 Jul 3;135(1):1-8. doi: 10.7326/0003-4819-135-1-200107030-00003. PMID 11434726
- [Background] Grodstein F, Manson JE, Colditz GA, Willett WC, Speizer FE, Stampfer MJ. A prospective, observational study of postmenopausal hormone therapy and primary prevention of cardiovascular disease. Ann Intern Med. 2000 Dec 19;133(12):933-41. doi: 10.7326/0003-4819-133-12-200012190-00008. PMID 11119394
- [Background] Hu FB, Bronner L, Willett WC, Stampfer MJ, Rexrode KM, Albert CM, Hunter D, Manson JE. Fish and omega-3 fatty acid intake and risk of coronary heart disease in women. JAMA. 2002 Apr 10;287(14):1815-21. doi: 10.1001/jama.287.14.1815. PMID 11939867
- [Background] Barr RG, Herbstman J, Speizer FE, Camargo CA Jr. Validation of self-reported chronic obstructive pulmonary disease in a cohort study of nurses. Am J Epidemiol. 2002 May 15;155(10):965-71. doi: 10.1093/aje/155.10.965. PMID 11994237
- [Background] Curhan GC, Willett WC, Rosner B, Stampfer MJ. Frequency of analgesic use and risk of hypertension in younger women. Arch Intern Med. 2002 Oct 28;162(19):2204-8. doi: 10.1001/archinte.162.19.2204. PMID 12390063
- [Background] Ayas NT, White DP, Al-Delaimy WK, Manson JE, Stampfer MJ, Speizer FE, Patel S, Hu FB. A prospective study of self-reported sleep duration and incident diabetes in women. Diabetes Care. 2003 Feb;26(2):380-4. doi: 10.2337/diacare.26.2.380. PMID 12547866
- [Background] Ayas NT, White DP, Manson JE, Stampfer MJ, Speizer FE, Malhotra A, Hu FB. A prospective study of sleep duration and coronary heart disease in women. Arch Intern Med. 2003 Jan 27;163(2):205-9. doi: 10.1001/archinte.163.2.205. PMID 12546611
- [Background] Albert CM, Chae CU, Grodstein F, Rose LM, Rexrode KM, Ruskin JN, Stampfer MJ, Manson JE. Prospective study of sudden cardiac death among women in the United States. Circulation. 2003 Apr 29;107(16):2096-101. doi: 10.1161/01.CIR.0000065223.21530.11. Epub 2003 Apr 14. PMID 12695299
- [Background] Knight EL, Stampfer MJ, Hankinson SE, Spiegelman D, Curhan GC. The impact of protein intake on renal function decline in women with normal renal function or mild renal insufficiency. Ann Intern Med. 2003 Mar 18;138(6):460-7. doi: 10.7326/0003-4819-138-6-200303180-00009. PMID 12639078
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Al-Delaimy WK, Mahoney GN, Speizer FE, Willett WC. Toenail nicotine levels as a biomarker of tobacco smoke exposure. Cancer Epidemiol Biomarkers Prev. 2002 Nov;11(11):1400-4. PMID 12433718
- [Background] Al-Delaimy WK, Manson JE, Willett WC, Stampfer MJ, Hu FB. Snoring as a risk factor for type II diabetes mellitus: a prospective study. Am J Epidemiol. 2002 Mar 1;155(5):387-93. doi: 10.1093/aje/155.5.387. PMID 11867347
- [Background] Feskanich D, Hastrup JL, Marshall JR, Colditz GA, Stampfer MJ, Willett WC, Kawachi I. Stress and suicide in the Nurses' Health Study. J Epidemiol Community Health. 2002 Feb;56(2):95-8. doi: 10.1136/jech.56.2.95. PMID 11812806
- [Background] Al-Delaimy WK, Willett WC, Manson JE, Speizer FE, Hu FB. Smoking and mortality among women with type 2 diabetes: The Nurses' Health Study cohort. Diabetes Care. 2001 Dec;24(12):2043-8. doi: 10.2337/diacare.24.12.2043. PMID 11723080
- [Background] Osganian SK, Stampfer MJ, Rimm E, Spiegelman D, Hu FB, Manson JE, Willett WC. Vitamin C and risk of coronary heart disease in women. J Am Coll Cardiol. 2003 Jul 16;42(2):246-52. doi: 10.1016/s0735-1097(03)00575-8. PMID 12875759
- [Background] Osganian SK, Stampfer MJ, Rimm E, Spiegelman D, Manson JE, Willett WC. Dietary carotenoids and risk of coronary artery disease in women. Am J Clin Nutr. 2003 Jun;77(6):1390-9. doi: 10.1093/ajcn/77.6.1390. PMID 12791615
- [Background] Jiang R, Hu FB, Giovannucci EL, Rimm EB, Stampfer MJ, Spiegelman D, Rosner BA, Willett WC. Joint association of alcohol and folate intake with risk of major chronic disease in women. Am J Epidemiol. 2003 Oct 15;158(8):760-71. doi: 10.1093/aje/kwg221. PMID 14561666
- [Background] Liu S, Willett WC, Manson JE, Hu FB, Rosner B, Colditz G. Relation between changes in intakes of dietary fiber and grain products and changes in weight and development of obesity among middle-aged women. Am J Clin Nutr. 2003 Nov;78(5):920-7. doi: 10.1093/ajcn/78.5.920. PMID 14594777
- [Background] Hu FB. Plant-based foods and prevention of cardiovascular disease: an overview. Am J Clin Nutr. 2003 Sep;78(3 Suppl):544S-551S. doi: 10.1093/ajcn/78.3.544S. PMID 12936948
- [Background] Knight EL, Stampfer MJ, Rimm EB, Hankinson SE, Curhan GC. Moderate alcohol intake and renal function decline in women: a prospective study. Nephrol Dial Transplant. 2003 Aug;18(8):1549-54. doi: 10.1093/ndt/gfg228. PMID 12897093
- [Background] Tanasescu M, Cho E, Manson JE, Hu FB. Dietary fat and cholesterol and the risk of cardiovascular disease among women with type 2 diabetes. Am J Clin Nutr. 2004 Jun;79(6):999-1005. doi: 10.1093/ajcn/79.6.999. PMID 15159229
- [Background] Cannuscio CC, Colditz GA, Rimm EB, Berkman LF, Jones CP, Kawachi I. Employment status, social ties, and caregivers' mental health. Soc Sci Med. 2004 Apr;58(7):1247-56. doi: 10.1016/S0277-9536(03)00317-4. PMID 14759673
- [Background] Mozaffarian D, Pischon T, Hankinson SE, Rifai N, Joshipura K, Willett WC, Rimm EB. Dietary intake of trans fatty acids and systemic inflammation in women. Am J Clin Nutr. 2004 Apr;79(4):606-12. doi: 10.1093/ajcn/79.4.606. PMID 15051604
- [Background] Rich-Edwards JW, Stampfer MJ, Manson JE, Rosner B, Hu FB, Michels KB, Willett WC. Breastfeeding during infancy and the risk of cardiovascular disease in adulthood. Epidemiology. 2004 Sep;15(5):550-6. doi: 10.1097/01.ede.0000129513.69321.ba. PMID 15308954
- [Background] Weinstein AR, Sesso HD, Lee IM, Cook NR, Manson JE, Buring JE, Gaziano JM. Relationship of physical activity vs body mass index with type 2 diabetes in women. JAMA. 2004 Sep 8;292(10):1188-94. doi: 10.1001/jama.292.10.1188. PMID 15353531
- [Background] Pai JK, Pischon T, Ma J, Manson JE, Hankinson SE, Joshipura K, Curhan GC, Rifai N, Cannuscio CC, Stampfer MJ, Rimm EB. Inflammatory markers and the risk of coronary heart disease in men and women. N Engl J Med. 2004 Dec 16;351(25):2599-610. doi: 10.1056/NEJMoa040967. PMID 15602020
- [Background] Oh K, Hu FB, Cho E, Rexrode KM, Stampfer MJ, Manson JE, Liu S, Willett WC. Carbohydrate intake, glycemic index, glycemic load, and dietary fiber in relation to risk of stroke in women. Am J Epidemiol. 2005 Jan 15;161(2):161-9. doi: 10.1093/aje/kwi026. PMID 15632266
- [Background] Hu FB, Willett WC, Li T, Stampfer MJ, Colditz GA, Manson JE. Adiposity as compared with physical activity in predicting mortality among women. N Engl J Med. 2004 Dec 23;351(26):2694-703. doi: 10.1056/NEJMoa042135. PMID 15616204
- [Background] Albert CM, Chae CU, Rexrode KM, Manson JE, Kawachi I. Phobic anxiety and risk of coronary heart disease and sudden cardiac death among women. Circulation. 2005 Feb 1;111(4):480-7. doi: 10.1161/01.CIR.0000153813.64165.5D. PMID 15687137
- [Background] Schulze MB, Shai I, Manson JE, Li T, Rifai N, Jiang R, Hu FB. Joint role of non-HDL cholesterol and glycated haemoglobin in predicting future coronary heart disease events among women with type 2 diabetes. Diabetologia. 2004 Dec;47(12):2129-36. doi: 10.1007/s00125-004-1593-2. Epub 2004 Dec 15. PMID 15662553
- [Background] Erkkila AT, Booth SL, Hu FB, Jacques PF, Manson JE, Rexrode KM, Stampfer MJ, Lichtenstein AH. Phylloquinone intake as a marker for coronary heart disease risk but not stroke in women. Eur J Clin Nutr. 2005 Feb;59(2):196-204. doi: 10.1038/sj.ejcn.1602058. PMID 15454972
- [Background] Al-Delaimy WK, Rexrode KM, Hu FB, Albert CM, Stampfer MJ, Willett WC, Manson JE. Folate intake and risk of stroke among women. Stroke. 2004 Jun;35(6):1259-63. doi: 10.1161/01.STR.0000127813.12854.9c. Epub 2004 Apr 22. PMID 15105514
- [Background] Forman JP, Rimm EB, Stampfer MJ, Curhan GC. Folate intake and the risk of incident hypertension among US women. JAMA. 2005 Jan 19;293(3):320-9. doi: 10.1001/jama.293.3.320. PMID 15657325
- [Background] Oh K, Hu FB, Manson JE, Stampfer MJ, Willett WC. Dietary fat intake and risk of coronary heart disease in women: 20 years of follow-up of the nurses' health study. Am J Epidemiol. 2005 Apr 1;161(7):672-9. doi: 10.1093/aje/kwi085. PMID 15781956
- [Background] Shai I, Schulze MB, Manson JE, Rexrode KM, Stampfer MJ, Mantzoros C, Hu FB. A prospective study of soluble tumor necrosis factor-alpha receptor II (sTNF-RII) and risk of coronary heart disease among women with type 2 diabetes. Diabetes Care. 2005 Jun;28(6):1376-82. doi: 10.2337/diacare.28.6.1376. PMID 15920055
- [Background] Mukamal KJ, Jensen MK, Gronbaek M, Stampfer MJ, Manson JE, Pischon T, Rimm EB. Drinking frequency, mediating biomarkers, and risk of myocardial infarction in women and men. Circulation. 2005 Sep 6;112(10):1406-13. doi: 10.1161/CIRCULATIONAHA.105.537704. Epub 2005 Aug 29. PMID 16129796
- [Background] Pai JK, Kraft P, Cannuscio CC, Manson JE, Rexrode KM, Albert CM, Hunter D, Rimm EB. Polymorphisms in the CC-chemokine receptor-2 (CCR2) and -5 (CCR5) genes and risk of coronary heart disease among US women. Atherosclerosis. 2006 May;186(1):132-9. doi: 10.1016/j.atherosclerosis.2005.06.041. Epub 2005 Aug 1. PMID 16055130
- [Background] Rich-Edwards JW, Kleinman K, Michels KB, Stampfer MJ, Manson JE, Rexrode KM, Hibert EN, Willett WC. Longitudinal study of birth weight and adult body mass index in predicting risk of coronary heart disease and stroke in women. BMJ. 2005 May 14;330(7500):1115. doi: 10.1136/bmj.38434.629630.E0. Epub 2005 Apr 27. PMID 15857857
- [Background] Albert CM, Oh K, Whang W, Manson JE, Chae CU, Stampfer MJ, Willett WC, Hu FB. Dietary alpha-linolenic acid intake and risk of sudden cardiac death and coronary heart disease. Circulation. 2005 Nov 22;112(21):3232-8. doi: 10.1161/CIRCULATIONAHA.105.572008. PMID 16301356
- [Background] Chiuve SE, Cook NR, Shay CM, Rexrode KM, Albert CM, Manson JE, Willett WC, Rimm EB. Lifestyle-based prediction model for the prevention of CVD: the Healthy Heart Score. J Am Heart Assoc. 2014 Nov 14;3(6):e000954. doi: 10.1161/JAHA.114.000954. PMID 25398889
- [Background] Qi Q, Kilpelainen TO, Downer MK, Tanaka T, Smith CE, Sluijs I, Sonestedt E, Chu AY, Renstrom F, Lin X, Angquist LH, Huang J, Liu Z, Li Y, Asif Ali M, Xu M, Ahluwalia TS, Boer JM, Chen P, Daimon M, Eriksson J, Perola M, Friedlander Y, Gao YT, Heppe DH, Holloway JW, Houston DK, Kanoni S, Kim YM, Laaksonen MA, Jaaskelainen T, Lee NR, Lehtimaki T, Lemaitre RN, Lu W, Luben RN, Manichaikul A, Mannisto S, Marques-Vidal P, Monda KL, Ngwa JS, Perusse L, van Rooij FJ, Xiang YB, Wen W, Wojczynski MK, Zhu J, Borecki IB, Bouchard C, Cai Q, Cooper C, Dedoussis GV, Deloukas P, Ferrucci L, Forouhi NG, Hansen T, Christiansen L, Hofman A, Johansson I, Jorgensen T, Karasawa S, Khaw KT, Kim MK, Kristiansson K, Li H, Lin X, Liu Y, Lohman KK, Long J, Mikkila V, Mozaffarian D, North K, Pedersen O, Raitakari O, Rissanen H, Tuomilehto J, van der Schouw YT, Uitterlinden AG, Zillikens MC, Franco OH, Shyong Tai E, Ou Shu X, Siscovick DS, Toft U, Verschuren WM, Vollenweider P, Wareham NJ, Witteman JC, Zheng W, Ridker PM, Kang JH, Liang L, Jensen MK, Curhan GC, Pasquale LR, Hunter DJ, Mohlke KL, Uusitupa M, Cupples LA, Rankinen T, Orho-Melander M, Wang T, Chasman DI, Franks PW, Sorensen TI, Hu FB, Loos RJ, Nettleton JA, Qi L. FTO genetic variants, dietary intake and body mass index: insights from 177,330 individuals. Hum Mol Genet. 2014 Dec 20;23(25):6961-72. doi: 10.1093/hmg/ddu411. Epub 2014 Aug 7. PMID 25104851
- [Background] Paik JM, Curhan GC, Sun Q, Rexrode KM, Manson JE, Rimm EB, Taylor EN. Calcium supplement intake and risk of cardiovascular disease in women. Osteoporos Int. 2014 Aug;25(8):2047-56. doi: 10.1007/s00198-014-2732-3. Epub 2014 May 7. PMID 24803331
- [Background] Sun Q, Jimenez MC, Townsend MK, Rimm EB, Manson JE, Albert CM, Rexrode KM. Plasma levels of fetuin-A and risk of coronary heart disease in US women: the Nurses' Health Study. J Am Heart Assoc. 2014 Jun 24;3(3):e000939. doi: 10.1161/JAHA.114.000939. PMID 24963103
- [Background] Yang S, Jensen MK, Rimm EB, Willett W, Wu T. Erythrocyte superoxide dismutase, glutathione peroxidase, and catalase activities and risk of coronary heart disease in generally healthy women: a prospective study. Am J Epidemiol. 2014 Nov 1;180(9):901-8. doi: 10.1093/aje/kwu195. Epub 2014 Aug 24. PMID 25156995
- [Background] Schnatz PF, Manson JE. Vitamin D and cardiovascular disease: an appraisal of the evidence. Clin Chem. 2014 Apr;60(4):600-9. doi: 10.1373/clinchem.2013.211037. Epub 2013 Nov 5. PMID 24193116
- [Background] Crous-Bou M, Fung TT, Prescott J, Julin B, Du M, Sun Q, Rexrode KM, Hu FB, De Vivo I. Mediterranean diet and telomere length in Nurses' Health Study: population based cohort study. BMJ. 2014 Dec 2;349:g6674. doi: 10.1136/bmj.g6674. PMID 25467028
- [Background] Mayers JR, Wu C, Clish CB, Kraft P, Torrence ME, Fiske BP, Yuan C, Bao Y, Townsend MK, Tworoger SS, Davidson SM, Papagiannakopoulos T, Yang A, Dayton TL, Ogino S, Stampfer MJ, Giovannucci EL, Qian ZR, Rubinson DA, Ma J, Sesso HD, Gaziano JM, Cochrane BB, Liu S, Wactawski-Wende J, Manson JE, Pollak MN, Kimmelman AC, Souza A, Pierce K, Wang TJ, Gerszten RE, Fuchs CS, Vander Heiden MG, Wolpin BM. Elevation of circulating branched-chain amino acids is an early event in human pancreatic adenocarcinoma development. Nat Med. 2014 Oct;20(10):1193-1198. doi: 10.1038/nm.3686. Epub 2014 Sep 28. PMID 25261994
- [Background] Bhupathiraju SN, Tobias DK, Malik VS, Pan A, Hruby A, Manson JE, Willett WC, Hu FB. Glycemic index, glycemic load, and risk of type 2 diabetes: results from 3 large US cohorts and an updated meta-analysis. Am J Clin Nutr. 2014 Jul;100(1):218-32. doi: 10.3945/ajcn.113.079533. Epub 2014 Apr 30. PMID 24787496
- [Background] Li Y, Wang DD, Chiuve SE, Manson JE, Willett WC, Hu FB, Qi L. Dietary phosphatidylcholine intake and type 2 diabetes in men and women. Diabetes Care. 2015 Feb;38(2):e13-4. doi: 10.2337/dc14-2093. No abstract available. PMID 25614692
- [Background] Huang T, Xu M, Lee A, Cho S, Qi L. Consumption of whole grains and cereal fiber and total and cause-specific mortality: prospective analysis of 367,442 individuals. BMC Med. 2015 Mar 24;13:59. doi: 10.1186/s12916-015-0294-7. PMID 25858689
- [Background] Li Y, Ley SH, Tobias DK, Chiuve SE, VanderWeele TJ, Rich-Edwards JW, Curhan GC, Willett WC, Manson JE, Hu FB, Qi L. Birth weight and later life adherence to unhealthy lifestyles in predicting type 2 diabetes: prospective cohort study. BMJ. 2015 Jul 21;351:h3672. doi: 10.1136/bmj.h3672. PMID 26199273
- [Background] Malik VS, Chiuve SE, Campos H, Rimm EB, Mozaffarian D, Hu FB, Sun Q. Circulating Very-Long-Chain Saturated Fatty Acids and Incident Coronary Heart Disease in US Men and Women. Circulation. 2015 Jul 28;132(4):260-8. doi: 10.1161/CIRCULATIONAHA.114.014911. Epub 2015 Jun 5. PMID 26048094
- [Background] Laugsand LE, Ix JH, Bartz TM, Djousse L, Kizer JR, Tracy RP, Dehghan A, Rexrode K, Lopez OL, Rimm EB, Siscovick DS, O'Donnell CJ, Newman A, Mukamal KJ, Jensen MK. Fetuin-A and risk of coronary heart disease: A Mendelian randomization analysis and a pooled analysis of AHSG genetic variants in 7 prospective studies. Atherosclerosis. 2015 Nov;243(1):44-52. doi: 10.1016/j.atherosclerosis.2015.08.031. Epub 2015 Sep 5. PMID 26343871
- [Background] Huang T, Zheng Y, Qi Q, Xu M, Ley SH, Li Y, Kang JH, Wiggs J, Pasquale LR, Chan AT, Rimm EB, Hunter DJ, Manson JE, Willett WC, Hu FB, Qi L. DNA Methylation Variants at HIF3A Locus, B-Vitamin Intake, and Long-term Weight Change: Gene-Diet Interactions in Two U.S. Cohorts. Diabetes. 2015 Sep;64(9):3146-54. doi: 10.2337/db15-0264. Epub 2015 May 22. PMID 26001398
- [Background] Li Y, Ley SH, VanderWeele TJ, Curhan GC, Rich-Edwards JW, Willett WC, Forman JP, Hu FB, Qi L. Joint association between birth weight at term and later life adherence to a healthy lifestyle with risk of hypertension: a prospective cohort study. BMC Med. 2015 Jul 31;13:175. doi: 10.1186/s12916-015-0409-1. PMID 26228391
- [Background] Chiuve SE, Sun Q, Sandhu RK, Tedrow U, Cook NR, Manson JE, Albert CM. Adiposity throughout adulthood and risk of sudden cardiac death in women. JACC Clin Electrophysiol. 2015 Dec 1;1(6):520-528. doi: 10.1016/j.jacep.2015.07.011. PMID 26824079
- [Background] Bassuk SS, Manson JE. Oral contraceptives and menopausal hormone therapy: relative and attributable risks of cardiovascular disease, cancer, and other health outcomes. Ann Epidemiol. 2015 Mar;25(3):193-200. doi: 10.1016/j.annepidem.2014.11.004. Epub 2014 Nov 13. PMID 25534509
- [Background] Garcia M, Mulvagh SL, Merz CN, Buring JE, Manson JE. Cardiovascular Disease in Women: Clinical Perspectives. Circ Res. 2016 Apr 15;118(8):1273-93. doi: 10.1161/CIRCRESAHA.116.307547. PMID 27081110
- [Background] Zheng Y, Li Y, Rimm EB, Hu FB, Albert CM, Rexrode KM, Manson JE, Qi L. Dietary phosphatidylcholine and risk of all-cause and cardiovascular-specific mortality among US women and men. Am J Clin Nutr. 2016 Jul;104(1):173-80. doi: 10.3945/ajcn.116.131771. Epub 2016 Jun 8. PMID 27281307
- [Background] Zheng Y, Xu M, Li Y, Hruby A, Rimm EB, Hu FB, Wirth J, Albert CM, Rexrode KM, Manson JE, Qi L. Gallstones and Risk of Coronary Heart Disease: Prospective Analysis of 270 000 Men and Women From 3 US Cohorts and Meta-Analysis. Arterioscler Thromb Vasc Biol. 2016 Sep;36(9):1997-2003. doi: 10.1161/ATVBAHA.116.307507. Epub 2016 Aug 18. PMID 27540264
- [Background] Yu E, Rimm E, Qi L, Rexrode K, Albert CM, Sun Q, Willett WC, Hu FB, Manson JE. Diet, Lifestyle, Biomarkers, Genetic Factors, and Risk of Cardiovascular Disease in the Nurses' Health Studies. Am J Public Health. 2016 Sep;106(9):1616-23. doi: 10.2105/AJPH.2016.303316. Epub 2016 Jul 26. PMID 27459449
- [Background] Chen M, Li Y, Sun Q, Pan A, Manson JE, Rexrode KM, Willett WC, Rimm EB, Hu FB. Dairy fat and risk of cardiovascular disease in 3 cohorts of US adults. Am J Clin Nutr. 2016 Nov;104(5):1209-1217. doi: 10.3945/ajcn.116.134460. Epub 2016 Aug 24. PMID 27557656
- [Background] Mora S, Manson JE. Aspirin for Primary Prevention of Atherosclerotic Cardiovascular Disease: Advances in Diagnosis and Treatment. JAMA Intern Med. 2016 Aug 1;176(8):1195-204. doi: 10.1001/jamainternmed.2016.2648. PMID 27322595
- [Background] Manson JE, Woodruff TK. Reproductive Health as a Marker of Subsequent Cardiovascular Disease: The Role of Estrogen. JAMA Cardiol. 2016 Oct 1;1(7):776-777. doi: 10.1001/jamacardio.2016.2662. No abstract available. PMID 27626902
- [Background] Ma W, Li Y, Heianza Y, Staller KD, Chan AT, Rimm EB, Rexrode KM, Qi L. Associations of Bowel Movement Frequency with Risk of Cardiovascular Disease and Mortality among US Women. Sci Rep. 2016 Sep 6;6:33005. doi: 10.1038/srep33005. PMID 27596972
- [Background] Bhupathiraju SN, Grodstein F, Stampfer MJ, Willett WC, Hu FB, Manson JE. Exogenous Hormone Use: Oral Contraceptives, Postmenopausal Hormone Therapy, and Health Outcomes in the Nurses' Health Study. Am J Public Health. 2016 Sep;106(9):1631-7. doi: 10.2105/AJPH.2016.303349. Epub 2016 Jul 26. PMID 27459451
- [Background] Hruby A, Manson JE, Qi L, Malik VS, Rimm EB, Sun Q, Willett WC, Hu FB. Determinants and Consequences of Obesity. Am J Public Health. 2016 Sep;106(9):1656-62. doi: 10.2105/AJPH.2016.303326. Epub 2016 Jul 26. PMID 27459460
- [Background] Manson JE, Kaunitz AM. Menopause Management--Getting Clinical Care Back on Track. N Engl J Med. 2016 Mar 3;374(9):803-6. doi: 10.1056/NEJMp1514242. No abstract available. PMID 26962899
- [Background] Legato MJ, Johnson PA, Manson JE. Consideration of Sex Differences in Medicine to Improve Health Care and Patient Outcomes. JAMA. 2016 Nov 8;316(18):1865-1866. doi: 10.1001/jama.2016.13995. No abstract available. PMID 27802499
- [Background] Wang T, Huang T, Kang JH, Zheng Y, Jensen MK, Wiggs JL, Pasquale LR, Fuchs CS, Campos H, Rimm EB, Willett WC, Hu FB, Qi L. Habitual coffee consumption and genetic predisposition to obesity: gene-diet interaction analyses in three US prospective studies. BMC Med. 2017 May 9;15(1):97. doi: 10.1186/s12916-017-0862-0. PMID 28486942
- [Background] Yu Z, Huang T, Zheng Y, Wang T, Heianza Y, Sun D, Campos H, Qi L. PCSK9 variant, long-chain n-3 PUFAs, and risk of nonfatal myocardial infarction in Costa Rican Hispanics. Am J Clin Nutr. 2017 May;105(5):1198-1203. doi: 10.3945/ajcn.116.148106. Epub 2017 Mar 22. PMID 28330911
- [Background] Ding M, Huang T, Bergholdt HK, Nordestgaard BG, Ellervik C, Qi L; CHARGE Consortium. Dairy consumption, systolic blood pressure, and risk of hypertension: Mendelian randomization study. BMJ. 2017 Mar 16;356:j1000. doi: 10.1136/bmj.j1000. PMID 28302601
- [Background] Heianza Y, Ma W, Manson JE, Rexrode KM, Qi L. Gut Microbiota Metabolites and Risk of Major Adverse Cardiovascular Disease Events and Death: A Systematic Review and Meta-Analysis of Prospective Studies. J Am Heart Assoc. 2017 Jun 29;6(7):e004947. doi: 10.1161/JAHA.116.004947. PMID 28663251
- [Derived] Liu X, Guasch-Ferre M, Drouin-Chartier JP, Tobias DK, Bhupathiraju SN, Rexrode KM, Willett WC, Sun Q, Li Y. Changes in Nut Consumption and Subsequent Cardiovascular Disease Risk Among US Men and Women: 3 Large Prospective Cohort Studies. J Am Heart Assoc. 2020 Apr 7;9(7):e013877. doi: 10.1161/JAHA.119.013877. Epub 2020 Apr 1. PMID 32233756
- [Derived] Zong G, Liu G, Willett WC, Wanders AJ, Alssema M, Zock PL, Hu FB, Sun Q. Associations Between Linoleic Acid Intake and Incident Type 2 Diabetes Among U.S. Men and Women. Diabetes Care. 2019 Aug;42(8):1406-1413. doi: 10.2337/dc19-0412. Epub 2019 Jun 10. PMID 31182488
- [Derived] Liu X, Li Y, Tobias DK, Wang DD, Manson JE, Willett WC, Hu FB. Changes in Types of Dietary Fats Influence Long-term Weight Change in US Women and Men. J Nutr. 2018 Nov 1;148(11):1821-1829. doi: 10.1093/jn/nxy183. PMID 30247611
- [Derived] Eckel N, Li Y, Kuxhaus O, Stefan N, Hu FB, Schulze MB. Transition from metabolic healthy to unhealthy phenotypes and association with cardiovascular disease risk across BMI categories in 90 257 women (the Nurses' Health Study): 30 year follow-up from a prospective cohort study. Lancet Diabetes Endocrinol. 2018 Sep;6(9):714-724. doi: 10.1016/S2213-8587(18)30137-2. Epub 2018 May 31. PMID 29859908
- [Derived] Zong G, Li Y, Sampson L, Dougherty LW, Willett WC, Wanders AJ, Alssema M, Zock PL, Hu FB, Sun Q. Monounsaturated fats from plant and animal sources in relation to risk of coronary heart disease among US men and women. Am J Clin Nutr. 2018 Mar 1;107(3):445-453. doi: 10.1093/ajcn/nqx004. PMID 29566185
- [Derived] McKeown NM, Dashti HS, Ma J, Haslam DE, Kiefte-de Jong JC, Smith CE, Tanaka T, Graff M, Lemaitre RN, Rybin D, Sonestedt E, Frazier-Wood AC, Mook-Kanamori DO, Li Y, Wang CA, Leermakers ETM, Mikkila V, Young KL, Mukamal KJ, Cupples LA, Schulz CA, Chen TA, Li-Gao R, Huang T, Oddy WH, Raitakari O, Rice K, Meigs JB, Ericson U, Steffen LM, Rosendaal FR, Hofman A, Kahonen M, Psaty BM, Brunkwall L, Uitterlinden AG, Viikari J, Siscovick DS, Seppala I, North KE, Mozaffarian D, Dupuis J, Orho-Melander M, Rich SS, de Mutsert R, Qi L, Pennell CE, Franco OH, Lehtimaki T, Herman MA. Sugar-sweetened beverage intake associations with fasting glucose and insulin concentrations are not modified by selected genetic variants in a ChREBP-FGF21 pathway: a meta-analysis. Diabetologia. 2018 Feb;61(2):317-330. doi: 10.1007/s00125-017-4475-0. Epub 2017 Nov 2. PMID 29098321
- [Derived] Korngold EC, Januzzi JL Jr, Gantzer ML, Moorthy MV, Cook NR, Albert CM. Amino-terminal pro-B-type natriuretic peptide and high-sensitivity C-reactive protein as predictors of sudden cardiac death among women. Circulation. 2009 Jun 9;119(22):2868-76. doi: 10.1161/CIRCULATIONAHA.108.832576. Epub 2009 May 26. PMID 19470888
- See also: Nurses' Health Study website — https://www.nurseshealthstudy.org/